CLINICAL TRIAL: NCT07097532
Title: Cutaneous Silent Period-Based Comparison of Dorsal Root Ganglion Pulsed Radiofrequency and Transforaminal Epidural Steroid Injection in Lumbar Radicular Pain
Brief Title: Cutaneous Silent Period-Based Comparison of DRG-PRF and TFESI in Lumbar Radicular Pain
Acronym: CSP-LRP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ahmet başarı (Other Government)
Responsible Party: Sponsor-Investigator, ahmet başarı, Pain Specialist, Kayseri City Hospital
Organization: Kayseri City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CSP-DRGPRF-TFESI-2025
Record Dates: First submitted 2025-07-25; First posted 2025-07-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Lumbar Radicular Pain; Spinal; Inhibition
Keywords: Cutaneous Silent Period; Lumbar Radicular Pain; Dorsal Root Ganglion Pulsed Radiofrequency; Transforaminal Epidural Eteroid Injection
MeSH Terms: conditions — Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model with three groups: two patient groups with lumbar radicular pain, randomized to receive either dorsal root ganglion pulsed radiofrequency (DRG-PRF) or transforaminal epidural steroid injection (TFESI), and one healthy control group undergoing cutaneous silent period (CSP) measurement only. Patients are randomly allocated to the intervention arms. Each group is evaluated independently, with no crossover or sequential interventions. CSP, pain, and disability outcomes are assessed at baseline and at follow-up time points for comparison.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor responsible for CSP measurements is blinded to group allocation. No other parties are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DRG-PRF Group (Experimental): Patients diagnosed with lumbar radicular pain underwent pulsed radiofrequency treatment targeting the dorsal root ganglion at the L4-5 or L5-S1 spinal levels under fluoroscopic guidance. The cutaneous silent period (CSP), pain intensity measured by the Numeric Rating Scale (NRS), and functional disability assessed by the Oswestry Disability Index (ODI) were evaluated before and after the intervention.
  Interventions: Procedure: Radiofrequency
- TFESI Group (Active Comparator): Patients diagnosed with lumbar radicular pain underwent transforaminal epidural steroid injections at the L4-5 or L5-S1 spinal levels under fluoroscopic guidance. The cutaneous silent period (CSP), pain intensity measured by the Numeric Rating Scale (NRS), and functional disability assessed by the Oswestry Disability Index (ODI) were evaluated before and after the intervention.
  Interventions: Procedure: Transforaminal Epidural Steroid Injection
- Healthy Control Group (No Intervention): Healthy individuals with no known spinal pathology or neuropathic pain underwent cutaneous silent period (CSP) evaluation for comparison purposes. No interventional procedures were performed in this group.

INTERVENTIONS:
Procedure: Radiofrequency — Under sterile conditions and fluoroscopic guidance, pulsed radiofrequency treatment was applied unilaterally to the dorsal root ganglia at the L4-L5 and L5-S1 spinal levels. Sensory and motor stimulation were performed to confirm appropriate electrode placement. Pulsed radiofrequency was delivered at 45 volts for 300 seconds at 42°C using standard radiofrequency equipment. Patients were monitored for three hours following the procedure, and cutaneous silent period (CSP) recordings were obtained on the same day and during follow-up assessments.
  Other Names: Dorsal Root Ganglion Radiofrequency
  Arms: DRG-PRF Group
Procedure: Transforaminal Epidural Steroid Injection — Using a fluoroscopic C-arm device, transforaminal epidural steroid injection (TFESI) was performed at the L4-L5 and L5-S1 foraminal levels. At each level, a total of 4 mL of solution containing 16 mg of dexamethasone and sterile saline was administered following confirmation of appropriate contrast spread. Negative aspiration was verified prior to injection. Cutaneous silent period (CSP) measurements were conducted on the same day and at designated follow-up intervals.
  Other Names: Transforaminal Epidural Steroid Injections
  Arms: TFESI Group

SUMMARY:
This prospective clinical study compares the effects of two interventional treatments, dorsal root ganglion pulsed radiofrequency (DRG-PRF) and transforaminal epidural steroid injection (TFESI), on patients with lumbar radicular pain (LRP). A third group of healthy individuals is included as a control group to provide baseline cutaneous silent period (CSP) values.

The CSP is a neurophysiological marker of spinal inhibition. The study aims to evaluate whether these treatments affect pain levels, functional disability, and CSP parameters over time. Participants with LRP will receive either DRG-PRF or TFESI, while healthy controls will undergo CSP testing only.

The findings may provide insight into the effects of these interventions on segmental nociceptive processing and inform treatment strategies for neuropathic low back pain.

DETAILED DESCRIPTION:
Lumbar radicular pain (LRP) is one of the most common causes of low back pain (1). It frequently results from disc herniation at the L4-5 or L5-S1 levels or from irritation of spinal nerve roots due to other degenerative conditions (2). Transforaminal epidural steroid injection (TFESI) and dorsal root ganglion pulsed radiofrequency (DRG-PRF) are minimally invasive interventional procedures used in the treatment of this condition. However, data objectively comparing the effects of these interventions on segmental nociceptive processing in humans are limited (3,4).

This prospective clinical study aims to evaluate both the clinical and neurophysiological effects of DRG-PRF and TFESI in individuals with LRP. The cutaneous silent period (CSP), a non-invasive electrophysiological marker that reflects spinal inhibitory function, will be used as an objective assessment tool. CSP is a polysynaptic spinal reflex in which a nociceptive stimulus conducted via A-delta fibers causes temporary suppression of voluntary motor activity (5). It represents the electrophysiological correlate of a protective reflex involving both sensory and motor pathways and enables functional assessment of thinly myelinated sensory fibers using standard neurophysiological equipment (6).

The study will include three groups: a DRG-PRF group, a TFESI group, and a healthy control group with no spinal pathology. Participants in the DRG-PRF and TFESI groups will be randomly allocated to treatment arms according to their order of presentation at the outpatient clinic. All participants will undergo baseline CSP recordings. In the treatment groups, CSP will be reassessed on Day 1, Week 1, and Month 1 following the intervention. CSP measurements will be conducted by an experienced electrophysiologist who is blinded to the treatment group. In addition, pain severity using the Numeric Rating Scale (NRS) and functional disability using the Oswestry Disability Index (ODI) will be evaluated in the treatment groups.

The DRG-PRF group will receive fluoroscopy-guided pulsed radiofrequency treatment at the L4-5 and L5-S1 lumbar levels using a standard 42°C protocol. The TFESI group will receive transforaminal corticosteroid injections at the same spinal levels. All procedures will be performed under sterile conditions by an experienced pain specialist.

The primary outcome of the study is to assess changes in CSP parameters, specifically onset latency and duration. Secondary outcomes include changes in pain intensity and functional capacity. The inclusion of a healthy control group will allow for comparison of CSP responses against normative values.

The study is expected to yield new insights into the neurophysiological effects of interventional pain treatments and to clarify the potential utility of CSP in monitoring treatment response in lumbar radicular pain. The findings may support more personalized clinical decision-making and enhance understanding of the underlying spinal mechanisms associated with these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Clinically and radiologically confirmed lumbar radicular pain (LRP) due to unilateral intervertebral disc herniation, confirmed by MRI and physical examination
* Symptom duration greater than 3 months
* Baseline pain score of ≥4 on the 11-point Numerical Rating Scale (NRS-11)
* Inadequate response to conservative treatment (e.g., medication or physical therapy)

Exclusion Criteria:

* Unstable or uncontrolled psychiatric illness
* Pregnancy
* Bleeding diathesis
* Known allergy to any procedural agent (e.g., local anesthetics, corticosteroids, contrast media)
* Prior lumbar surgery
* Spondylolisthesis
* Compression fracture
* Discitis
* Bilateral or sequestered disc herniation
* Moderate-to-severe spinal stenosis
* Diabetes mellitus
* Polyneuropathy
* Fibromyalgia
* Movement disorders
* Regular use of antidepressants or tramadol
* Regular use of pregabalin or gabapentin
* Chronic alcohol use
* Noncompliance with follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-07-08 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
Change in Cutaneous Silent Period (CSP) Parameters | Baseline, Day 1, Week 1, and Month 1 post-procedure
  Evaluation of changes in electrophysiological parameters of the cutaneous silent period (CSP), including onset latency, offset latency, and duration, recorded from the tibialis anterior muscle following sural nerve stimulation. These parameters are used to assess segmental spinal inhibitory function and to evaluate the modulatory effects of dorsal root ganglion pulsed radiofrequency (DRG-PRF) and transforaminal epidural steroid injection (TFESI) in patients with lumbar radicular pain.

SECONDARY OUTCOMES:
Change in Clinical Outcomes: Pain Intensity and Functional Disability | Baseline, Day 1, Week 1, and Month 1 post-procedure
  Clinical outcomes will be assessed using the 11-point Numerical Rating Scale (NRS-11) for pain intensity and the Oswestry Disability Index (ODI) for functional disability. NRS-11 scores will be measured at baseline, day 1, week 1, and month 1, while ODI scores will be evaluated at baseline and month 1. These measures will be used to determine the clinical effectiveness of dorsal root ganglion pulsed radiofrequency (DRG-PRF) and transforaminal epidural steroid injection (TFESI) in patients with lumbar radicular pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Basari, Pain Specialist, Neurologist, Principal Investigator — Kayseri City Hospital
Locations (1):
- Kayseri City Hospital, Kayseri, Seker, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared due to institutional data protection policy and ethical constraints.

REFERENCES:
- [Background] Kofler M, Leis AA, Valls-Sole J. Cutaneous silent periods - Part 1: Update on physiological mechanisms. Clin Neurophysiol. 2019 Apr;130(4):588-603. doi: 10.1016/j.clinph.2019.01.002. Epub 2019 Jan 18. PMID 30691969
- [Background] Floeter MK. Cutaneous silent periods. Muscle Nerve. 2003 Oct;28(4):391-401. doi: 10.1002/mus.10447. PMID 14506711
- [Background] Gunduz OH, Sencan S, Ercalik T, Suhaimi A. Recovery of H-Reflex with Transforaminal Epidural Steroid Injection in S1 Radiculopathy. Pain Med. 2017 Aug 1;18(8):1594-1597. doi: 10.1093/pm/pnw303. No abstract available. PMID 28087843
- [Background] Vigneri S, Sindaco G, La Grua M, Zanella M, Paci V, Vinci FM, Sciacca C, Merlini A, Pari G. Long-term Inhibition of Soleus H-reflex with Epidural Adhesiolysis and Pulsed Radiofrequency in Lumbosacral Neuropathic Pain. Pain Pract. 2021 Mar;21(3):277-284. doi: 10.1111/papr.12955. Epub 2020 Oct 25. PMID 32970918
- [Background] Van Boxem K, Cheng J, Patijn J, van Kleef M, Lataster A, Mekhail N, Van Zundert J. 11. Lumbosacral radicular pain. Pain Pract. 2010 Jul-Aug;10(4):339-58. doi: 10.1111/j.1533-2500.2010.00370.x. Epub 2010 May 17. PMID 20492580
- [Background] Manchikanti L, Singh V, Falco FJ, Benyamin RM, Hirsch JA. Epidemiology of low back pain in adults. Neuromodulation. 2014 Oct;17 Suppl 2:3-10. doi: 10.1111/ner.12018. PMID 25395111